CLINICAL TRIAL: NCT06534476
Title: The Effect of Education Given to Hemodialysis Patients on Patients' Self-Care Ability and Fluid Control
Brief Title: Effectiveness of Education Given to Patients With Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Yildirim (Other)
Responsible Party: Sponsor-Investigator, Zeynep Yildirim, PhD Student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZeynepY
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Nurse's Role
Keywords: Hemodialysis; Patient Education; Self-Care Ability; Fluid Control
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education (Experimental): The intervention group was given 40-50 minutes of training.
  Interventions: Other: Education
- Control Group (No Intervention): Routine nursing care was given to hemodialysis patients in this group without any training.

INTERVENTIONS:
Other: Education — Patients who agreed to participate in the study and met the inclusion criteria were interviewed face to face before the HD session and their verbal and written permissions were obtained by reading the voluntary consent form. The researcher interviewed the patients one-on-one and provided information about the purpose of the study and the training program. Then, scale forms were applied to the patients. In order not to interrupt the training and not to distract the patients in this group, a separate room in the Dialysis Unit was used during the training. The education booklet "Living with Hemodialysis" on hemodialysis management prepared in line with the literature was given to the patients by the researcher. The training of a patient lasted an average of 40-50 minutes. During and at the end of the training, the patients' questions were answered in the training room.
  Arms: Patient Education

SUMMARY:
This study was conducted to investigate the effects of education given to patients receiving hemodialysis treatment on self-care agency and fluid control. This study has a pre-test-post-test quasi-experimental design. A total of 54 hemodialysis patients who met the inclusion criteria were included in the study.

DETAILED DESCRIPTION:
Chronic diseases are one of the major public health problems. Chronic renal failure (CKD) is among the chronic diseases that cause death worldwide. CKD is defined as a chronic and progressive deterioration in the kidney's fluid-solute balance adjustment and metabolic-endocrine functions resulting from a decrease in glomerular filtration rate. CKD affects approximately 10-15% of adults worldwide and 15.7% of adults in Turkey. Renal replacement treatment options for CKD are peritoneal dialysis, hemodialysis (HD) and kidney transplantation. The most common treatment method applied is HD. It was reported that 76% of patients with CKD in Turkey at the end of 2017 received HD treatment. The aim of HD is to correct the patient's fluid and electrolyte imbalance, prevent possible complications, compensate for the patient's lost renal functions as much as possible and increase the quality of life. However, in addition to these, diet causes negativities such as fluid restriction, depression, job loss, loss of role in family life, fear of death, and decreased self-care ability in HD patients. Self-care ability is defined as "a dynamic process that enables individuals to participate in health services". Lack of self-care ability makes it difficult to adapt to the disease. Therefore, it negatively affects the treatment and increases the cost of the disease. Self-care behaviors in HD patients include appropriate diet intake, regular medication use, compliance with fluid restriction, and coping with stress. Studies show that there is a correlation between the level of self-care in HD patients and compliance with treatment, health-enhancing behaviors, and the reduction of physical and psychological symptoms. For this reason, it is important to develop self-care ability in order to protect and improve the quality of life of HD patients and to prevent possible complications. The area that creates the most stress in HD and makes it difficult to comply with treatment is fluid restriction. Non-compliance with fluid restriction is reported as 30.6-95% in Turkey and 15.3-80% worldwide. As the disease progresses, HD patients lose their ability to form urine. Therefore, the amount of fluid consumed becomes important. In addition, excessive fluid loading in patients increases mortality rates. For this reason, fluid restriction control should be made a lifestyle in disease management. Nurses who respond to and intervene in patients' needs instantly have great duties and responsibilities. It can be said that nursing care and education are of great importance in solving existing or potential problems of individuals receiving HD treatment. Patient education, which is within the scope of the nurse's educational role, ensures that the patient is protected from possible complications, can control fluids, increases self-care ability, and gains behavioral changes related to their health. The effects of education given to HD patients on various parameters have been examined in the literature. However, no study examining the self-care ability and fluid restriction of education has been found. Therefore, this study was conducted to examine the effects of education given to patients receiving HD treatment on self-care ability and fluid control.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old and above
* Receiving dialysis treatment for at least three months
* Being literate

Exclusion Criteria:

* Having communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Self-Care Ability Scale | Up to 8 weeks
  Self-care ability scale, developed by Besey Ören in 2010, consists of 22 items and five sub-dimensions. These dimensions are; drug use (1, 2, 3, 4, 5, 18), diet (8, 9, 10, 11, 12), hygienic care (15, 16, 17, 19), mental state (20, 21, 22) and self-monitoring (6,7,13, 14). The scale is a 3-point Likert type (0: I never apply, 1: I sometimes apply, 2: I always apply). Items 12, 20, 21, 22 on the scale are scored negatively. The scores obtained from the scale range from 0 to 44. According to the scale, as the scores obtained increase, the self-care ability of patients receiving dialysis treatment increases.
Fluid Control Scale in Hemodialysis Patients | Up to 8 weeks
  Fluid control scale in hemodialysis patients, developed by Coşar and Çınar in 2012 consists of 24 items and three sub-dimensions. These sub-dimensions are; knowledge (1-7), behavior (8-18) and attitude (19-24). The scale is a 3-point Likert type (1: Disagree, 2: Undecided, 3: Agree). Items 7, 18, 19, 20, 21, 22, 23 and 24 in the scale are scored negatively. Scores obtained from the scale range from 24 to 72. As the score obtained increases, the patients' compliance with fluid control increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No